CLINICAL TRIAL: NCT00003694
Title: A Phase II Study of Newly Diagnosed Patients With BCR/ABL (+) Chronic Myelogenous Leukemia Treated With Combined Homoharringtonine (NSC #141633) and Low-Dose Cytarabine
Brief Title: Homoharringtonine Plus Low-Dose Cytarabine in Treating Patients With Newly Diagnosed Chronic Myelogenous Leukemia in Chronic Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02786; CALGB-19804; U10CA031946 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-12-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Homoharringtonine; Cytarabine

ARMS (1):
- Treatment (omacetaxine mepesuccinate, cytarabine) (Experimental): Patients receive cytarabine and homoharringtonine concurrently by continuous intravenous infusion for 7 days. Courses repeat every 28 days. Patients receive a minimum of 9 courses of therapy in the absence of disease progression and unacceptable toxicity. Patients who are major cytogenetic responders at 9 months may continue therapy or switch to interferon. Minor cytogenetic responders are switched to interferon, and nonresponders are removed from therapy and given the option to switch to interferon.
  Interventions: Drug: omacetaxine mepesuccinate; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: omacetaxine mepesuccinate — Given IV
  Other Names: CGX-635; homoharringtonine
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of homoharringtonine plus low-dose cytarabine in treating patients who have newly diagnosed chronic phase chronic myelogenous leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the hematologic and cytogenetic response rate of newly diagnosed patients with BCR/ABL (+) chronic myelogenous leukemia (CML) treated with combined homoharringtonine (omacetaxine mepesuccinate) and low dose cytarabine.

II. To estimate the toxicity of these two drugs given in combination in a cooperative group setting.

SECONDARY OBJECTIVES:

I. To assess duration of hematological response and incidence of hematological progression for all patients.

II. To assess duration of cytogenetic response in patients continuing protocol therapy beyond the initial nine months.

III. To use quantitative Southern blot monitoring of blood samples to monitor molecular response rates in patients entered onto CALGB treatment studies for CML.

IV. To compare quantitative Southern blot results of blood samples with marrow cytogenetics at the time of complete molecular response.

V. To use RT-PCR to monitor the frequency of residual disease in patients who have achieved a complete blood Southern blot and marrow cytogenetic response (elimination of BCR/ABL positivity by Southern blot and absence of the Philadelphia chromosome by cytogenetics).

OUTLINE:

Patients receive cytarabine and homoharringtonine concurrently by continuous intravenous infusion for 7 days. Courses repeat every 28 days. Patients receive a minimum of 9 courses of therapy in the absence of disease progression and unacceptable toxicity. Patients who are major cytogenetic responders at 9 months may continue therapy or switch to interferon. Minor cytogenetic responders are switched to interferon, and nonresponders are removed from therapy and given the option to switch to interferon.

Patients are followed every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of chronic myelogenous leukemia (CML) in chronic phase; patients in either accelerated or blastic phases are not eligible; clonal cytogenetic evolution alone does not exclude patients
* Patients must meet one or more of the following criteria:

  * Cytogenetically determined Philadelphia chromosome (Ph+)
  * BCR/ABL protein detectable by immunoblotting
  * Polymerase chain reaction (PCR) positive fusion transcripts for BCR/ABL
  * BCR/ABL translocation present by fluorescence in situ hybridization (FISH)
* Registration within eight weeks of the diagnosis and confirmation of Ph+ or BCR/ABL+ CML
* No more than eight weeks of prior hydroxyurea therapy
* No previous therapy with homoharringtonine (HHT)
* No prior treatment for CML with agents other than hydroxyurea; thus, prior treatment for CML with agents such as interferon, busulfan or cytarabine will render patients ineligible
* Must not be a candidate for an early allogeneic bone marrow transplant; potential transplant candidates must be counseled about alternative donor transplants and must decline that treatment option
* ECOG performance status 0-2
* Non-pregnant and non-nursing; treatment under this protocol would expose an unborn child to significant risks; women and men of reproductive potential should agree to use an effective means of birth control
* Bilirubin =< x upper limit of normal
* Creatinine =< 1.5 mg/dl

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1999-03; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Complete cytogenetic, major cytogenetic, and hematologic response rate | Up to 9 months
  Two separate single-stage Fleming designs will be used to test hypotheses regarding the major cytogenetic response rate and the complete cytogenetic response rate. Calculated and presented with their 95% confidence intervals.

SECONDARY OUTCOMES:
Toxicity rates as assessed by Common Terminology Criterial version 2.0 | Up to 9 months
Duration of hematological response | Up to 10 years
  Described with Kaplan-Meier curves.
Time to hematological progression | Up to 10 years
  Described with Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Dana-Farber Harvard Cancer Center, Boston, Massachusetts, United States